CLINICAL TRIAL: NCT03082924
Title: Surface Diaphragm EMG Evaluate the Clinical Efficacy of Pulmonary Rehabilitation in Patients With Chronic Obstructive Pulmonary Disease: a Multi Center Prospective Randomized Controlled Study
Brief Title: Surface EMGdi Evaluate the Efficacy of Pulmonary Rehabilitation in Patients With COPD: a Multi Center Prospective Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhujiang Hospital (Other)
Collaborators: Guangzhou Institute of Respiratory Disease (Other); The First Affiliated Hospital of Guangdong Pharmaceutical University (Other); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CX20160902
Record Dates: First submitted 2016-12-27; First posted 2017-03-17 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2017-03

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: surface EMGdi; pulmonary rehabilitation; inspiratory muscle training; exercise training
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Control group (Experimental): Neither cycle training nor inspiratory muscle training.
  Interventions: Device: Control group
- Cycle training group (Experimental): A calibrated cycle ergometer is used to do 30-minute cycling training session 3 days a week.
  Interventions: Device: Calibrated cycle ergometer
- Inspiratory training group (Experimental): A threshold loading device is used to perform 21-minute inspiratory muscle training 3 days a week.
  Interventions: Device: Threshold loading device
- Combined group (Experimental): Calibrated cycle ergometer and threshold loading device are applied.A 30-minute cycle training is performed using calibrated cycle ergometer and a 21-minute inspiratory muscle training using threshold loading device 3 days a week.
  Interventions: Device: Calibrated cycle ergometer and threshold loading device

INTERVENTIONS:
Device: Control group — Neither cycle training nor inspiratory muscle training.
  Arms: Control group
Device: Calibrated cycle ergometer — The most common device to perform cycle training is calibrated cycle ergometer.
  Arms: Cycle training group
Device: Threshold loading device — Threshold loading device is used to perform inspiratory muscle training.
  Arms: Inspiratory training group
Device: Calibrated cycle ergometer and threshold loading device — Combined cycle training and inspiratory muscle training.The threshold loading device is composed of a mouth -piece attached to a small plastic cylinder that contains a spring-loaded poppet value. The valve opens to permit inspiratory flow only once the person has generated adequate negative intrathoracic pressure to condense the spring.
  Arms: Combined group

SUMMARY:
Pulmonary rehabilitation is recognized as a core component of the management of individuals with chronic obstructive respiratory disease, which has become first-line treatment besides drug therapy. However, in the current clinical evaluation system of pulmonary rehabilitation, there is still a lack of simple, objective index,which can be monitored at any time.Neural respiratory drive , as an important physiological index, is closely related to the symptoms and the severity of the disease. It may be a sensitive indicator to evaluate the effectiveness of pulmonary rehabilitation. Surface EMGdi can accurately evaluate neural respiratory drive , its detection is non-invasive, simple and safety . In recent years, with the development of signal detection and analysis technology, EMG recording is more stable, but as the related research samples were low, surface diaphragm EMG has not yet the establishment of standardization. Therefore, based on the previous work, the project was carried out in a multicenter randomized controlled study,in which the stable stage of COPD patients were included in different ways of pulmonary rehabilitation training, a comprehensive clinical assessment will be conducted before and after training. Compared with the traditional evaluation methods and standard esophageal diaphragmatic electromyography, surface EMGdi detect the changes of neural respiratory drive in patients with COPD,that can help to explore the application value of surface EMGdi in the assessment of chronic obstructive pulmonary disease with pulmonary rehabilitation, to provide a basis for the promotion of the diaphragm and the optimization of pulmonary rehabilitation program.

DETAILED DESCRIPTION:
The patients with COPD will participate in a rehabilitation program for 52 weeks.

Participants in the proposed study will be randomly programmed into one of four intervention groups:

1. Neither cycle training nor inspiratory muscle training.
2. Cycle training program alone (performing on calibrated stationary cycle ergometer).
3. Inspiratory muscle training alone (performing on threshold loading device).
4. Combined cycle training and inspiratory muscle training(performing on calibrated stationary cycle ergometer and threshold loading device).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged over 40 years old.
* Patients with pulmonary function test of forced expiratory volume at one second(FEV1)/forced vital capacity(FVC) < 70%.
* Patients in a clinically stable state
* Patients who signed informed consent.
* No participation in other pulmonary rehabilitation program within the previous 2 months.

Exclusion Criteria:

* Patients with signs of an airway infection.
* Patients with metabolic disease and serious cardiovascular disease.
* Patients with Multiple pulmonary bulla.
* Patients with poor compliance.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2016-07; Primary Completion 2020-12 (Actual); Study Completion 2021-06 (Actual)

PRIMARY OUTCOMES:
Diaphragmatic function(composite outcome measure) | Change from baseline in diaphragm electromyogram.(8 weeks later, 26 weeks later, 52 weeks later)
  Diaphragmatic function can be assessed by diaphragm electromyogram (EMGdi), which reflect the physiological activity of the diaphragm and indicate functional status of the central drive.

SECONDARY OUTCOMES:
Inspiratory muscle function(composite outcome measure) | Change from baseline in inspiratory muscle function.(8 weeks later, 26 weeks later, 52 weeks later)
  Currently, the maximal inspiratory pressure (PImax) and maximal expiratory pressures(PEmax) are measured by a digital manometer (AZ-8205, AZ Instrument, Taichung City, Taiwan)and combined to evaluate inspiratory muscle function.
Pulmonary Function(composite outcome measure) | Change from baseline in pulmonary function.(8 weeks later, 26 weeks later, 52 weeks later)
  Pulmonary function is measured using a spirometer(PonyFX 229, Cosmed, Rome, Italy) that is calibrated daily.The FEV1 and percent-of-predicted FEV1, FVC and percent-of-predicted FVC which are presented in one report are used to evaluate Pulmonary Function.
Cardiopulmonary exercise test(composite outcome measure) | Change from baseline in cardiopulmonary exercise test.(8 weeks later, 26 weeks later, 52 weeks later)
  Cardiopulmonary exercise test can help to reflect the variables,like maximaloxygen uptake（VO2max）, anaerobic threshold (AT).
Degree of dyspnea(composite outcome measure) | Change from baseline in degree of dyspnea.(8 weeks later, 26 weeks later, 52 weeks later)
  Difference in the degree of dyspnea can be measured by Borg index.
Exercise capacity(composite outcome measure) | Change from baseline in exercise performance.(8 weeks later, 26 weeks later, 52 weeks later)
  Exercise capacity is evaluated using the 6-min walking distance (6MWD) according to American Thoracic Society guidelines.

OTHER OUTCOMES:
Body Composition Monitor(composite outcome measure) | Change from baseline in body composition.(8 weeks later, 26 weeks later, 52 weeks later)
  Body composition abnormalities are prevalent in COPD.Human body composition analyzer can detect various elements of human body and analyze human health status.
Health-related quality(composite outcome measure) | Change from baseline in Health-related quality.(8 weeks later, 26 weeks later, 52 weeks later)
  Health-related quality is a component of the broader concept of quality of life and is defined as satisfaction with health.The St. George's Respiratory Questionnaire (SGRQ) and Chronic Respiratory Disease Questionnaire (CRQ）;and its self-reported version are the most widely used disease-specific questionnaires.
Symptom Evaluation(composite outcome measure) | Change from baseline in symptom evaluation.(8 weeks later, 26 weeks later, 52 weeks later)
  Individuals with chronic respiratory disease often have symptoms such as dyspnea, fatigue, cough, weakness,sleeplessness,and psychological distress.Instruments for assessment of multiple symptoms include COPD Assessment Test (CAT) and Modified Medical British Research Council Scale(mMRC).
Depression and anxiety evaluation(composite outcome measure) | Change from baseline in depression and anxiety evaluatione.(8 weeks later, 26 weeks later, 52 weeks later)
  Hospital Anxiety and Depression Scale (HADS) was found to perform well in assessing the symptom severity and caseness of anxiety disorders and depression in both somatic, psychiatric and primary care patients and in the general population.

CONTACTS AND LOCATIONS:
Overall Officials: Xin Chen, Doctor, Principal Investigator — Zhujiang Hospital,Southern Medical Unversity
Locations (1):
- Zhujiang Hospital,Southern Medical Universtiy, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided